CLINICAL TRIAL: NCT06912373
Title: Experiences, Outcomes and Unmet Needs of Caregivers of Children With Cerebral Palsy in Spain: A Mixed-Method Study
Brief Title: Experiences, Outcomes and Unmet Needs of Caregivers of Children With Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Clàudia Arumí, Clàudia Arumí-Trujillo, Universitat de Lleida
Other Study IDs: ULleida3
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy Infantile; Caregiver
Keywords: Caregivers; Cerebral Palsy; Mixed-Method Research; Quality of Life; Parenting Stress
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cerebral Palsy caregivers: Quantitative data will be collected and analysed using three questionnaires, providing the authors with a comprehensive profile of participants' stress levels, quality of life, and caregiver burden. This data will also enable the identification of specific subgroups that will be the primary focus of the subsequent qualitative phase, while informing the development of new research questions for a deeper exploration during this phase. Participants who meet the inclusion criteria and have signed the informed consent will be directed to a study homepage hosted on the university's website. This website will provide a link to REDCap (Research Electronic Data Capture), a secure platform specifically designed for collecting research data (PedsQL-FIM, ZBI, PSS-14).

SUMMARY:
Cerebral palsy (CP ) is one of the most prevalent motor disabilities in childhood, significantly impacting both children and their caregivers. This study explores the experiences, psychological well-being, and unmet needs of caregivers of children with CP. Using an explanatory sequential design (QUAN → QUAL), first it will be assessed burden, stress levels, and quality of life of caregivers through standardized questionnaires (PedsQL-FIM , ZBI , PSS-14 ).

DETAILED DESCRIPTION:
Before the recruitment begins, the principal investigator will present the project to the pediatric service of the Arnau de Vilanova University Hospital of Lleida (HUAV). During medical consultations, the pediatric service will inform eligible participants about the study. If the caregiver agrees to participate, they will give consent for the pediatric service to share their contact details with the research team. The investigators will then contact the participant to explain the project in detail, schedule a first meeting to sign the Informed Consent, and complete the initial questionnaires. The Informed Consent will include the first author's contact information so that participants can address any questions or concerns about the study. Additionally, participants who sign the informed consent will be asked to provide their contact information for potential follow-up regarding the qualitative interview.

In the first meeting, participants who meet the inclusion criteria and have signed the informed consent will be directed to a study homepage hosted on the university's website. This website will provide a link to REDCap (Research Electronic Data Capture), a secure platform specifically designed for collecting research data (PedsQL-FIM, ZBI, PSS-14).

Participants' sociodemographic data will include descriptive information such as age, sex, household income, among others

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Being a caregiver of a child with Cerebral Palsy
* Spanish/Catalan speaking
* Willing to talk about their experiences and be audio/video-recorded.
* Accept and sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children with developmental disorders or disabilities. The birth of a child with cerebral palsy can significantly alter the family's daily life, leading parents to feel denial, sadness, and guilt. They need to adapt to their child's limitations and find ways to handle these new challenges. In this sense, the birth of a child diagnosed with a chronic illness or disability, has the potential to change the family routine, triggering feelings of denial, sadness and guilt in the parental figures who need to learn to face the limitations of their children .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Stress | Day 1
  The PSS-14 is short and easy adaptation of the original Perceived Stress Scale (PSS), with the original author being Cohen, S. The European Spanish adaptation was conducted by Remor, E.
  The PSS measures the degree to which individuals perceive life situations as stressful over the past month, focusing on subjective control over unpredictable events and the distress associated with perceived lack of control. The PSS is more closely related to subjective evaluations of life events than objective measures of stressors (18). The PSS-14 European Spanish version will be used and consists of 14 items scored from 0 up to 4 (0=never, 1 = rarely 2= sometimes 3= usually 4 =almost always). The total scores on the scale can range from 0 (no stress) to 56 (extreme stress). The European Spanish version PSS (14-item) demonstrated adequate reliability (internal consistency, alpha = .81, and test-retest, r = .73), validity (concurrent), and sensitivity

SECONDARY OUTCOMES:
The Quality of Life | Day 1
  To assess the impact of pediatric chronic health conditions on caregivers and the family, the Spanish version of the PedsQL™ Family Impact Module will be used. This module employs a multidimensional parent self-report to evaluate physical, emotional, social, and cognitive functioning, as well as communication and worry. The module can be completed within 5-10 minutes
  The PedsQL-FIM It is a 36-item with an internal consistency reliability of α = 0.97 (21). It assesses 8 main factors: physical functioning (6 items), emotional functioning (5 items), social functioning (4 items), cognitive functioning (4 items), communication (3 items), worry (5 items), daily activities (3 items) and family relationships (5 items). The answers are given on a 5-point Likert scale (0 = it is never a problem, 4 = it is almost always a problem) and are reversed scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). A greater score indicates better functioning.
Burden | Day 1
  To asses caregiver burden, the Zarit Burden Interview will be used. The Zarit Burden Interview is a widely used self-report instrument for measuring caregiver burden. ZBI assesses caregivers´ perceptions of burden that may inadvertently affect their health, personal, social or financial wellbeing.
  Caregivers are requested to assess the level of burden they experience while caring for a loved one. Burden is defined as the degree to which a caregiver perceives negative effects on their emotional and physical health, social life, and finances, which may hinder their ability to provide care. Responses vary from "not at all" to "extremely." It consists of 22 items, with the total score calculated by summing the scores of all the indicated items. It is suggested that a score from 0 to 21 means no to mild burden, 21 to 40 indicates mild to moderate burden, 41 to 60 indicates moderate to severe burden, and more than 61 means severe burden.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Valenzuela, PhD, Study Director — Universitat de Lleida

IPD SHARING:
Plan to Share IPD: No